CLINICAL TRIAL: NCT01417312
Title: Metabolic Effects of a Green Tea Extract in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Friedemann Paul, Prof, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MS_GTE
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple sclerosis; Green tea extract; Metabolism
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green tea extract (Active Comparator)
  Interventions: Dietary Supplement: Capsules with 160 mg Teavigo (at least 94% EGCG)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Capsules with 160 mg Teavigo (at least 94% EGCG) — Daily intake of 600 mg EGCG for 3 months
  Arms: Green tea extract
Dietary Supplement: Placebo — Daily intake of placebo capsules for 3 months
  Arms: Placebo

SUMMARY:
This study aims to investigate metabolic effects of a standardized green tea extract, containing a defined amount of epigallocatechin-3-gallate (EGCG), in multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing-remitting multiple sclerosis
* stable treatment with glatiramer acetate at least 6 months prior to inclusion
* Expanded disability status scale < 4.5
* Normal weight, overweight

Exclusion Criteria:

* Primary or secondary progressive forms of multiple sclerosis
* Clinically relevant heart, lung, liver, kidney diseases
* Habitual caffeine intake over 300 mg per day
* Habitual consumption of green tea
* Alcohol or drug abuse

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial lipid oxidation in grams per hour, assessed by indirect calorimetry, after 3 months intake of green tea extract versus placebo | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Prof, MD, Principal Investigator — NeuroCure Clinical Research Center and Experimental and Clinical Research Center, Charité University Medicine Berlin and Max Delbrueck Center for Molecular Medicine, Berlin, Germany; Michael Boschmann, MD, Principal Investigator — Franz-Volhard Clinical Research Center at the Experimental and Clinical Research Center, Charité University Medicine and Max Delbrueck Center for Molecular Medicine, Berlin, Germany
Locations (1):
- Franz-Volhard Clinical Research Center at the Experimental and Clinical Research Center, Charité University Medicine Berlin and Max Delbrueck Center for Molecular Medicine, Berlin, Germany

REFERENCES:
- [Derived] Mahler A, Steiniger J, Bock M, Klug L, Parreidt N, Lorenz M, Zimmermann BF, Krannich A, Paul F, Boschmann M. Metabolic response to epigallocatechin-3-gallate in relapsing-remitting multiple sclerosis: a randomized clinical trial. Am J Clin Nutr. 2015 Mar;101(3):487-95. doi: 10.3945/ajcn.113.075309. Epub 2015 Jan 14. PMID 25733633